CLINICAL TRIAL: NCT02706782
Title: An Open-label, Uncontrolled, Single-arm Pilot Study to Evaluate Vascular Interventional Therapy Mediated Mesothelin-targeted Chimeric Antigen Receptor T Cells in Advanced Pancreatic Carcinoma
Brief Title: A Study of Mesothelin Redirected Autologous T Cells for Advanced Pancreatic Carcinoma
Acronym: meso-CART
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai GeneChem Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Genechem meso-CART
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAI-meso-CART (Experimental): A single dose of meso-CART cells will be administered by vascular interventional mediated as one dose infusions. The dose is 1-10x106/kg meso-CAR positive T cells. The infusion will be scheduled to occur 2 days after a single dose of 1.5 grams/m2 of cyclophosphamide, which will be administered according to standard procedures. Patients will undergo cannula--DSA radiography--CAR-T cells perfusion. The cells perfusion process would lasts 15min to 2 h, and the specific time depends on patent's tumor-burdened state.
  Interventions: Drug: TAI-meso-CART

INTERVENTIONS:
Drug: TAI-meso-CART — TAI as a local drug delivery pathway, so that more T cells gathered at the tumor site, less T cells to migrate to the normal tissue, thereby enhancing the efficacy of anti-tumor, reducing the potential of side effects. And meso-CART is a 2nd CAR, with mesothelin as target protein, 4-1BB as co- stimulator
  Other Names: Transcatheter Arterial Infusion of meso-CART cells

SUMMARY:
Pancreatic carcinoma typically has a high recurrence rate and very poor prognosis. Surgery is the best choice for the treatment of pancreatic cancer, but for those advanced pancreatic cancer patients，when surgery is not available，chemotherapy combined with radiation therapy or interventional therapy is commonly used in the treatment，but the prolonging survival effect is not obvious. And now, some clinical researchers use CAR-T cells in the treatment of pancreatic carcinoma, according to the existing results, therapeutic effects are not as good as expecting. One of the most likely reasons is that they continued to use the intravenous infusing of CART cells to patients, when the T cells into the blood circulation, will result in decreased tumor activity and more potential adverse effects. We believe that a suitable TAA targeted-CAR-T cells will be an effective way to treat cancer, as long as the pathway of the cell infused to the body can not only improve the drug concentration of the tumor site but reduce the potential off-target side effects. In order to achieve this goal, it is probably the best choice to use vascular intervention to mediate CAR-T cells infusion. Mesothelin is a cell-surface antigen implicated in tumor invasion, which is highly expressed in pancreatic carcinoma but low-level expressed in mesothelia. We design a 2nd CART cells targeted with mesothelin, and use vascular intervention mediated CAR-T infusion to patients. We hope deliver anti-mesothelin CART cells locally can reducing the side effects while enhancing the antitumor affect by more CART cells accumulate in tumor sites while less can reach normal mesothelial tissue.

DETAILED DESCRIPTION:
This study is being conducted to assess vascular interventional therapy mediated anti-mesothelin-CAR-T(meso-CAR-T) cells safety and efficacy in treating patients with advanced pancreatic carcinoma.The investigators constructed a 2nd CAR, using mesothelin as target, using 4-1BB as co-stimulator. The source of T cells used to prepare CAR-T should be autologous. The infusion dose is (1-10)×106 meso-CAR positive T cells/kg, and the specific cells numbers depends on the situation of individual CAR-T cells preparation. The infusion way is vascular interventional mediated, which would undergo cannula--DSA radiography--CAR-T cells perfusion. The cells perfusion process would lasts 15min to 2 h, and the specific time depends on patent's tumor-burdened state.

ELIGIBILITY:
Inclusion Criteria:

* Mesothelin expression positive and histologically confirmed as pancreatic carcinoma;
* Aged between 18 and 69;
* Persistent cancer after at least one prior standard of care chemotherapy, has no willing for surgery or cannot be suitable for surgery patients with or without liver, lymph node metastasis;
* Tumor is too big to surgical resection;
* Life expectancy greater than 4 months;
* Satisfactory organ and bone marrow function as defined by the following: (1) creatinine <1.5mg/dl; (2) albumin >2; (3) cardiac ejection fraction of >55%; (4) ALT/AST<3×the institution normal upper limit; (5) hemoglobin>9g/dl, bilirubin 2.0×the institution normal upper limit; (6) absolute neutrophil count >1,000/ul, platelets>75,000/ul;
* Without bleeding disorder or coagulation disorders;
* Don't allergy to radiocontrast agent;
* Birth control;
* Adequate venous access for apheresis, and no other contraindications for leukapheresis;
* Voluntary informed consent is given.

Exclusion Criteria:

* Pregnant or lactating women;
* Uncontrolled active infection;
* Active hepatitis B or hepatitis C infection;
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary;
* Previously treatment with any gene therapy products;
* Feasibility assessment during screening demonstrates<30% transduction of target lymphocytes, or insufficient expansion (<5-fold) in response to CD3/CD28 costimulation;
* Any serious, uncontrolled diseases (including, but not limit to, unstable angina pectoris, congestive heart failure, grade III or IV cardiac disease, serious arrhythmia, liver and kidney disorders or metabolic diseases, CNS diseases).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-02 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse event | 6 weeks
  asverse event is evaluated with CTCAE, version 4.0

SECONDARY OUTCOMES:
Number of patients with tumor response | 8 weeks
  summarize tumor response by overal response rates
Detection of transferred T cells in the circulation using quantitative -PCR | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu Aimin, Doctor, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided